CLINICAL TRIAL: NCT01115179
Title: Propofol and/or Its Solvent Modify the Course of Inflammatory Response After Surgical Stress: A Randomized, Controlled, Double-blind Study
Brief Title: Propofol and Perioperative Inflammation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Bara Ricou, Service of Intensive Care, Department APSI, Geneva University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: APSIC 04-014; CER: 04-189 (Other: Ethics Comission)
Record Dates: First submitted 2010-04-27; First posted 2010-05-04 (Estimated); Last update posted 2010-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Inflammation
Keywords: propofol; inflammation; perioperative; lipids; Apolipoprotein A-I
MeSH Terms: conditions — Inflammation | interventions — Propofol; soybean oil, phospholipid emulsion; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Propofol (Active Comparator): Propofol anesthesia
  Interventions: Drug: propofol
- Control (Active Comparator): Anesthesia with isoflurane alone
  Interventions: Drug: Saline
- Solvent (Active Comparator): Anesthesia with isoflurane together with the solvent of propofol (intralipid)
  Interventions: Drug: Intralipid 10%

INTERVENTIONS:
Drug: propofol — Induction with propofol (1.5 to 2mg/kg) and maintenance of anesthesia with propofol 1% (target controlled infusion with concentration levels of 3-5 ug/ml)
  Other Names: Propofol, Ansiven
  Arms: Propofol
Drug: Intralipid 10% — Induction of anesthesia with thiopental (3-5mg/kg) and maintenance of anesthesia with isoflurane (end-expired concentration = 0.5%-2.0%) as well as the solvent of propofol 1% (Intralipid 10%; corresponding to a target-controlled infusion of propofol with concentration levels of 3-5ug/ml)
  Other Names: Intralipid
  Arms: Solvent
Drug: Saline — Induction of anesthesia with thiopental (3-5mg/kg) and maintenance of anesthesia with isoflurane (end-expired concentration = 0.5%-2.0%)
  Other Names: NaCl 0.9%
  Arms: Control

SUMMARY:
The inflammatory properties of propofol are still under debate. Apolipoprotein A-I (Apo A-I) is involved in the inflammatory process. This study was designed to determine whether and how propofol or its solvent modulate Apo A-I and the inflammatory response after surgical stress. The investigators study hypothesis was that propofol might modify the Apo A-I blood levels, and thus, modulate the postoperative inflammatory course.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I or II
* scheduled for uni- or bilateral elective laparoscopic totally extraperitoneal hernia repair

Exclusion Criteria:

* Body mass index (BMI) < 18.5 or > 39.9kg/m2
* treatments with steroids (>5mg/d prednisone equivalent, for the last 30 days)
* with opioids/non-steroidal anti-inflammatory drugs (NSAIDs) for chronic pain during the last 30 days
* immunosuppression (AIDS, neutropenia <1000 cells/ml, transplant surgery, chemotherapy)
* known lipid disorder (triglycerides >2.00mmol/l, low-density lipoprotein (LDL)-cholesterol >2.50mmol/l or high-density lipoprotein (HDL)-cholesterol < 1.00mmol/l)
* hypolipemic treatment before admission
* thyroid metabolism disorder (thyroid-stimulating hormone >6.0 mUI/l or <0.4mUI/l)
* renal insufficiency (creatinine >106umol/l)
* liver disorder (bilirubin >20umol/l, thromboplastin time <60%)
* insulin dependant diabetes
* parenteral nutrition or after any lipid-containing medication (propofol, intralipid, etomidate) during the last 30 days
* antihypertensive medication with diltiazem or other calcium channel blockers
* known chronic alcoholism (men: >65-75 ml alcohol/day)
* multidrug abuse (cocaine, heroin, methadone, or other narcotics, sedatives or stimulants)
* mental illness
* known allergy to propofol after randomization:
* change of surgical strategy
* protocol violation
* major bleeding (>0.5l)

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2005-03; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Apolipoprotein A-I level | 24 hours after surgery

SECONDARY OUTCOMES:
Interleukin-6 level | 5 hours after surgery
C-reactive protein (CRP) level | 24 hours after surgery
Cortisol level | 15 min after induction of anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Bara Ricou, Prof., Study Chair — Service of Intensive Care, Geneva University Hospital; Oliver Bandschapp, M.D., Principal Investigator — Service of Intensive Care, Geneva University Hospital
Locations (1):
- Service of Anesthesiology; Geneva University Hospital, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Background] Chenaud C, Merlani PG, Roux-Lombard P, Burger D, Harbarth S, Luyasu S, Graf JD, Dayer JM, Ricou B. Low apolipoprotein A-I level at intensive care unit admission and systemic inflammatory response syndrome exacerbation. Crit Care Med. 2004 Mar;32(3):632-7. doi: 10.1097/01.ccm.0000114820.47460.0a. PMID 15090939
- [Background] Hyka N, Dayer JM, Modoux C, Kohno T, Edwards CK 3rd, Roux-Lombard P, Burger D. Apolipoprotein A-I inhibits the production of interleukin-1beta and tumor necrosis factor-alpha by blocking contact-mediated activation of monocytes by T lymphocytes. Blood. 2001 Apr 15;97(8):2381-9. doi: 10.1182/blood.v97.8.2381. PMID 11290601